CLINICAL TRIAL: NCT05236322
Title: Management of Plasma Cell Gingivitis by En-block Removal
Brief Title: Management of Plasma Cell Gingivitis by Two Surgical Techniques
Acronym: PCG
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, principle investigator, Ain Shams University
Other Study IDs: 1232022
Record Dates: First submitted 2022-01-23; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Plasma Cell Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The sample and will be examined to ensure the final diagnosis of lesion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Removal by soft tissue laser of the tumor
  Interventions: Device: soft tissue laser
- control group: Removal by ordinary surgical scalpel

INTERVENTIONS:
Device: soft tissue laser — Surgical laser used in excision purpose
  Groups: study group

SUMMARY:
Two surgical protocols for management of Plasma cell Ginigivitis; either by surgical enblock resection of cold laser resection

DETAILED DESCRIPTION:
Tow groups will be included the first will have six cases and second will have six cases. the first will be treated by ordinary surgical resection and second will be removed using soft tissue laser.

ELIGIBILITY:
Inclusion Criteria:

- patients suffering from the plasma cell gingivitis

Exclusion Criteria:

- Patient not eligible for maxillofacial surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient suffering from plasma cell gingivitis
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
complete removal | one month
  complete removal of lesion with safety margin

CONTACTS AND LOCATIONS:
Overall Officials: mohamed diaa, professor, Study Chair — Ain Shams University
Locations (1):
- Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
yes planning to share